CLINICAL TRIAL: NCT00316602
Title: A Multicenter, Open-label, Controlled Phase II Study to Evaluate Immunogenicity and Safety of MVA-BN® (IMVAMUNE™) Smallpox Vaccine in 18-40 Year Old Subjects With Diagnosed Atopic Dermatitis
Brief Title: A Phase II Study on Immunogenicity and Safety of MVA-BN® (IMVAMUNE™) Smallpox Vaccine in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: POX-MVA-008; HHSN266200400072C (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2006-04-20; First posted 2006-04-21 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Smallpox; Vaccination
MeSH Terms: conditions — Dermatitis, Atopic; Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Participants (Experimental): Healthy, vaccinia naive subjects without Atopic Dermatitis, receiving two doses of MVA-BN (IMVAMUNE)
  Interventions: Biological: IMVAMUNE
- Atopic Dermatitis Participants (Experimental): Vaccinia naive subjects with diagnosed Atopic Dermatitis. "Diagnosed" AD included subjects with either history of or subjects with currently active AD (defined as scoring AD [SCORAD] <= 30), receiving two doses of MVA-BN (IMVAMUNE)
  Interventions: Biological: IMVAMUNE

INTERVENTIONS:
Biological: IMVAMUNE — Subjects receiving two subcutaneous vaccinations
  Other Names: MVA-BN

SUMMARY:
The purpose of this study is to compare the immunogenicity and safety of an investigational smallpox vaccine in subjects with atopic dermatitis to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (Healthy Participants):

Subjects without present or history of any kind of atopy.

Group 2 (Atopic Dermatitis Participants):

Subjects with diagnosed atopic dermatitis.

All study subjects:

1. Male and female subjects between 18 and 40 years of age without history of smallpox vaccination.
2. Women must have a negative serum pregnancy test at screening and a negative urine or serum pregnancy test within 24 hours prior to vaccination.
3. Women of childbearing potential must have used an acceptable method of contraception for 30 days prior to the first vaccination, must agree to use an acceptable method of contraception during the study, and must not become pregnant for at least 28 days after the last vaccination.
4. Lab values without clinically significant findings.
5. Electrocardiogram (ECG) without clinically significant findings.

Exclusion Criteria:

1. Pregnant or breast-feeding women.
2. Uncontrolled serious infection i.e. not responding to antimicrobial therapy.
3. History of or active autoimmune disease. Persons with vitiligo or thyroid disease taking thyroid replacement are not excluded.
4. Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease; diabetes mellitus; moderate to severe kidney impairment.
5. History of malignancy, other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure. Subjects with history of skin cancer at the vaccination site are excluded.
6. History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure.
7. History of an immediate family member (father, mother, brother, or sister) who has had onset of ischemic heart disease before age 50 years.
8. Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool: (http://hin.nhlbi.nih.gov/atpiii/calculator.asp?usertype=prof) NOTE: This criterion applies only to volunteers 20 years of age and older.
9. History of anaphylaxis or severe allergic reaction.
10. Post organ transplant subjects whether or not receiving chronic immunosuppressive therapy.
11. Administration of immunomodulatory substances.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 632 (Actual)
Dates: Start 2006-07; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard N Greenberg, M.D., Principal Investigator — University of Kentucky School of Medicine
Locations (22):
- United States (15):
  - Alta Clinical Research LLC, Tucson, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Rx Clinical Research, Inc., Garden Grove, California
  - Solano Clinical Research, Vallejo, California
  - Northwestern University, Chicago, Illinois
  - Adult & Pediatric Dermatology PC, Overland Park, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Saint Louis University, St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Dermatology Associates of Rochester, Rochester, New York
  - Oregon Dermatology & Research Center, Portland, Oregon
  - Dermatology Treatment & Research Center, Dallas, Texas
  - Dermatology Clinical Research, San Antonio, Texas
- Mexico (7):
  - Hospital Juárez de México, Magdalena de las Salinas, CP
  - Instituto Dermatologico de Jalisco "Dr. Jose Barba Rubio", Guadalajara, Jalisco
  - Hospital General de México, Mexico City
  - CIFBIOTEC (Centro de Investigacion Farmacologica y Biotecnologica), Mexico City
  - Hospital Regional Lic. Adolfo Lopez Mateos. ISSSTE Ciudad de Mexico, Mexico City
  - Centro Regional de Alergia e Inmunología Clínica del Hospital Universitario "Dr. José Eleuterio González", Monterrey
  - Hospital Angel Leañol, Dermatology, Zapopan, Jalisco

REFERENCES:
- [Result] Greenberg RN, Hurley MY, Dinh DV, Mraz S, Vera JG, von Bredow D, von Krempelhuber A, Roesch S, Virgin G, Arndtz-Wiedemann N, Meyer TP, Schmidt D, Nichols R, Young P, Chaplin P. A Multicenter, Open-Label, Controlled Phase II Study to Evaluate Safety and Immunogenicity of MVA Smallpox Vaccine (IMVAMUNE) in 18-40 Year Old Subjects with Diagnosed Atopic Dermatitis. PLoS One. 2015 Oct 6;10(10):e0138348. doi: 10.1371/journal.pone.0138348. eCollection 2015. PMID 26439129

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
Started | 282 | 350
Completed | 272 | 325
Not Completed | 10 | 25
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Subject unwilling/unable to comply with | 3 | 17
Not completed — Adverse Event | 1 | 0
Not completed — Other | 3 | 6

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Atopic Dermatitis Participants: Vaccinia naïve subjects with diagnosed AD. "Diagnosed" AD included subjects with either history of or subjects with currently active AD (defined as scoring AD [SCORAD] ≤ 30)
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Atopic Dermatitis Participants | Total
Number analyzed (Participants) | 282 | 350 | 632
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (5.81) | 27.9 (6.33) | 27.7 (6.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 223 | 373
  Male | 132 | 127 | 259
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 24 | 33 | 57
  Caucasian | 124 | 125 | 249
  Hispanic | 109 | 134 | 243
  Oriental/Asian | 20 | 49 | 69
  Other | 5 | 9 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 194 | 243 | 437
  Mexico | 88 | 107 | 195

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroconversion by ELISA
Description: Seroconversion rate based on Enzyme-linked Immunosorbent Assay (ELISA). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (50) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: week 6
Population: Per Protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
Number analyzed (Participants) | 194 | 257
percentage of subjects | 98.5 [95.5 to 99.7] | 97.3 [94.5 to 98.9]
Statistical Analysis 1: Comparison: Healthy Participants vs Atopic Dermatitis Participants; Test type: Non-Inferiority — The non-inferiority margin to show that Group 2 (Atopic Dermatitis Participants) is non-inferior to Group 1 (Healthy Participants) in terms of seroconversion rate at Week 6 was predefined as -5% for the difference in seroconversion rates; Difference in seroconversion rates (%) = -1.2, 97.5% CI 1-sided [lower limit -4.3]

2. Secondary Outcome: Percentage of Participants With Seroconversion by ELISA
Description: as for outcome 1
Time Frame: within 32 weeks
Population: Per Protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
Number analyzed (Participants) | 194 | 257
percentage of subjects
  Week 1: number analyzed (Participants) | 184 | 249
  Week 1 | 12.5 [8.1 to 18.2] | 22.9 [17.8 to 28.6]
  Week 4: number analyzed (Participants) | 192 | 254
  Week 4 | 85.4 [79.6 to 90.1] | 85.4 [80.5 to 89.5]
  Week 6 | 98.5 [95.5 to 99.7] | 97.3 [94.5 to 98.9]
  Week 8: number analyzed (Participants) | 188 | 244
  Week 8 | 98.4 [95.4 to 99.7] | 97.1 [94.2 to 98.8]
  Week 32: number analyzed (Participants) | 94 | 76
  Week 32 | 68.1 [57.7 to 77.3] | 75.0 [63.7 to 84.2]

3. Secondary Outcome: ELISA GMT
Description: Geometric Mean Titers (GMT) based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Titers below the detection limit are included with a value of '1'.
Time Frame: within 32 weeks
Population: Per Protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
Number analyzed (Participants) | 194 | 257
Titer
  Week 0 | 1.4 [1.2 to 1.7] | 1.7 [1.4 to 2.0]
  Week 1 | 2.2 [1.7 to 2.9] | 3.4 [2.6 to 4.4]
  Week 4 | 60.0 [47.2 to 76.4] | 62.3 [50.1 to 77.4]
  Week 6 | 499.4 [417.1 to 598.0] | 532.9 [452.9 to 627.1]
  Week 8 | 298.0 [252.3 to 351.8] | 314.3 [269.2 to 366.8]
  Week 32 | 21.4 [14.2 to 32.3] | 33.2 [21.7 to 50.6]

4. Secondary Outcome: Percentage of Participants With Seroconversion by PRNT
Description: Seroconversion rate based on Plaque Reduction Neutralization Test (PRNT). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (15) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: within 32 weeks
Population: Per Protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
Number analyzed (Participants) | 194 | 257
percentage of subjects
  Week 1: number analyzed (Participants) | 184 | 249
  Week 1 | 5.4 [2.6 to 9.8] | 5.6 [3.1 to 9.3]
  Week 4: number analyzed (Participants) | 192 | 254
  Week 4 | 24.5 [18.6 to 31.2] | 26.8 [21.4 to 32.7]
  Week 6 | 86.6 [81.0 to 91.1] | 90.3 [86.0 to 93.6]
  Week 8: number analyzed (Participants) | 188 | 244
  Week 8 | 76.1 [69.3 to 82.0] | 80.7 [75.2 to 85.5]
  Week 32: number analyzed (Participants) | 94 | 76
  Week 32 | 22.3 [14.4 to 32.1] | 19.7 [11.5 to 30.5]

5. Secondary Outcome: PRNT GMT
Description: Geometric Mean Titers (GMT) based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Titers below the detection limit are included with a value of '1'.
Time Frame: within 32 weeks
Population: Per Protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
Number analyzed (Participants) | 194 | 257
Titer
  Week 0 | 1.1 [1.0 to 1.2] | 1.2 [1.1 to 1.4]
  Week 1 | 1.3 [1.1 to 1.5] | 1.5 [1.2 to 1.7]
  Week 4 | 2.4 [1.9 to 3.1] | 2.8 [2.2 to 3.5]
  Week 6 | 34.6 [26.4 to 45.3] | 47.7 [38.1 to 59.8]
  Week 8 | 15.7 [12.0 to 20.6] | 21.9 [17.2 to 27.9]
  Week 32 | 2.2 [1.6 to 2.9] | 2.3 [1.6 to 3.5]

6. Secondary Outcome: ELISPOT IFN-γ Values
Description: Number of interferon gamma (IFN-γ) secreting peripheral blood mononuclear cells (PBMC) per 10^6 PBMC in response to restimulation with MVA-BN detected by ELISPOT assay
Time Frame: within 6 weeks
Population: ELISPOT Analysis Set
Measure: Median (Full Range); unit: Spot Forming Units / 10^6 PBMC
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
Number analyzed (Participants) | 46 | 71
Spot Forming Units / 10^6 PBMC
  Week 0 | 107.5 [0 to 775] | 109.0 [0 to 871]
  Week 1 | 106.5 [0 to 674] | 166.0 [0 to 1800]
  Week 6 | 276.5 [0 to 1800] | 334.0 [0 to 1800]

7. Secondary Outcome: Number of Participants With SAEs
Description: Occurrence, relationship and intensity of any serious AE (SAE)
Time Frame: within 32 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
Number analyzed (Participants) | 282 | 350
Participants
  Any SAE | 3 | 3
  Any SAE with intensity >= Grade 3 | 3 | 2
  Any SAE assessed as related to vaccine | 1 | 0

8. Secondary Outcome: Number of Participants With Related Grade >=3 Adverse Events
Description: Number of Participants with any Grade >=3 Adverse Event probably, possibly, or definitely related to the study vaccine. Pooled solicited (general) and unsolicited AEs.
Time Frame: within 29 days after vaccination
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
Number analyzed (Participants) | 282 | 350
Participants | 16 | 27

9. Secondary Outcome: Number of Participants With Solicited Local Adverse Events
Description: Number of Participants with and Intensity of solicited local AEs (erythema, swelling and pain). Percentages based on subjects with at least one completed diary card.
Time Frame: within 8 days after any vaccination
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
Number analyzed (Participants) | 282 | 345
Participants
  Pain : Total | 233 | 283
  Pain : Grade >=2 | 117 | 152
  Pain : Grade >=3 | 31 | 53
  Erythema : Total | 139 | 211
  Erythema : Grade >=2 | 35 | 66
  Erythema : Grade >=3 | 3 | 3
  Swelling : Total | 115 | 180
  Swelling : Grade >=2 | 21 | 45
  Swelling : Grade >=3 | 2 | 1

10. Secondary Outcome: Number of Participants With Solicited General AEs
Description: Number of Participants with solicited systemic/general AEs (elevated body temperature, headache, myalgia, nausea, fatigue and chills): Intensity and relationship to vaccination. Percentages based on subjects with at least one completed diary card.
Time Frame: within 8 days after any vaccination
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
Number analyzed (Participants) | 282 | 345
Participants
  Body Temperature increased : Total | 23 | 28
  Body Temperature increased : Related | 16 | 20
  Body Temperature increased : Grade >=3 | 1 | 1
  Body Temperature increased : Related - Grade >=3 | 1 | 1
  Headache : Total | 98 | 163
  Headache : Related | 76 | 119
  Headache : Grade >=3 | 9 | 26
  Headache : Related - Grade >=3 | 5 | 18
  Myalgia : Total | 98 | 153
  Myalgia : Related | 88 | 121
  Myalgia : Grade >=3 | 9 | 14
  Myalgia : Related - Grade >=3 | 8 | 9
  Chills : Total | 22 | 55
  Chills : Related | 19 | 39
  Chills : Grade >=3 | 4 | 7
  Chills : Related - Grade >=3 | 4 | 3
  Nausea : Total | 41 | 80
  Nausea : Related | 29 | 49
  Nausea : Grade >=3 | 6 | 8
  Nausea : Related - Grade >=3 | 4 | 5
  Fatigue : Total | 75 | 124
  Fatigue : Related | 53 | 90
  Fatigue : Grade >=3 | 9 | 16
  Fatigue : Related - Grade >=3 | 5 | 9

11. Secondary Outcome: Number of Unsolicited Non-serious Adverse Events: Intensity
Description: Occurrence of unsolicited non-serious AEs by Intensity
Time Frame: within 29 days after any vaccination
Population: Safety Analysis Set
Measure: Number; unit: events
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
Number analyzed (Participants) | 282 | 350
events
  Total | 432 | 538
  Grade 1 | 298 | 432
  Grade 2 | 108 | 86
  Grade 3 | 26 | 20
  Grade 4 | 0 | 0
  Missing | 0 | 0

12. Secondary Outcome: Number of Unsolicited Non-serious Adverse Events: Relationship to Vaccination
Description: Occurrence of unsolicited non-serious AEs by relationship to study vaccine
Time Frame: within 29 days after any vaccination
Population: Safety Analysis Set
Measure: Number; unit: events
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
Number analyzed (Participants) | 282 | 350
events
  None | 142 | 170
  Unlikely | 117 | 86
  Possible | 76 | 111
  Probable | 59 | 92
  Definite | 38 | 79
  Total | 432 | 538

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | Healthy Participants | Atopic Dermatitis Participants
All-Cause Mortality (participants affected / at risk) | 0/282 | 0/350
Serious Adverse Events (participants affected / at risk) | 3/282 | 3/350
Other Adverse Events (participants affected / at risk) | 133/282 | 196/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants (N=282) | Atopic Dermatitis Participants (N=350)
Extraocular muscle paresis (Eye disorders) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Loss of consciousness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Neurosis (Psychiatric disorders) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Participants (N=282) | Atopic Dermatitis Participants (N=350)
Injection site pruritus (General disorders) | 48 | 100
Injection site bruising (General disorders) | 2 | 7
Injection site induration (General disorders) | 6 | 3
Troponin I increased (Investigations) | 37 | 54
Nasopharyngitis (Infections and infestations) | 11 | 23
Influenza (Infections and infestations) | 8 | 11
Upper respiratory tract infection (Infections and infestations) | 9 | 6
Pharyngitis (Infections and infestations) | 9 | 4
Pharyngotonsillitis (Infections and infestations) | 7 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 9
Headache (Nervous system disorders) | 19 | 16
Dizziness (Nervous system disorders) | 7 | 11
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 7 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes